CLINICAL TRIAL: NCT06269978
Title: A Phase I Study of Intraperitoneal 5FU+Oxaliplatin in Patients With Colorectal Cancer With Isolated Peritoneal Metastasis
Brief Title: Intraperitoneal Oxaliplatin and Fluorouracil for the Treatment of Patients With Peritoneal Metastases From Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Arjun Mittra (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Arjun Mittra, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-23195; NCI-2023-10497 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R21CA282536 (NIH)
Record Dates: First submitted 2024-01-09; First posted 2024-02-21 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Colorectal Carcinoma; Metastatic Malignant Neoplasm in the Peritoneum; Stage IV Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Biopsy; Specimen Handling; Laparoscopy; Fluorouracil; dehydroftorafur; Magnetic Resonance Spectroscopy; Oxaliplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (oxaliplatin, 5FU) (Experimental): Patients undergo placement of indwelling IP port for chemotherapy infusion. Patients receive oxaliplatin and 5FU over 1-2 hours via IP infusion on days 1 and 15 of each cycle. Cycles repeat every 4 weeks for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo diagnostic laparoscopy, biopsy, CT/MRI, and collection of blood samples at screening and on study and undergo collection of IP fluid samples on study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Diagnostic Laparoscopy; Drug: Fluorouracil; Procedure: Magnetic Resonance Imaging; Drug: Oxaliplatin; Procedure: Surgical Procedure

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood and IP fluid samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Diagnostic Laparoscopy — Undergo diagnostic laparoscopy
Drug: Fluorouracil — Given via IP infusion
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Oxaliplatin — Given via IP infusion
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Procedure: Surgical Procedure — Undergo placement of indwelling IP port
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of intraperitoneal oxaliplatin and fluorouracil in treating patients with colorectal cancer that has spread to the peritoneal cavity (peritoneal metastasis). Oxaliplatin is in a class of medications called platinum-containing antineoplastic agents. It damages the cell's DNA and may kill cancer cells. Fluorouracil stops cells from making DNA and it may kill cancer cells. Both oxaliplatin and fluorouracil are approved by the Food and Drug Administration to treat patients with colorectal cancer, however administration of these drugs directly into the area between the muscles and organs in the abdomen (intraperitoneal) for the treatment of peritoneal metastases is experimental. Giving oxaliplatin and fluorouracil directly into the peritoneal space may be a safe and effective way of treating patients with peritoneal metastases from colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine safety, tolerability, and maximally tolerated dose (MTD) of intraperitoneal (IP) fluorouracil (5FU)+oxaliplatin.

II. Determine pharmacokinetics (PK) of IP 5FU+oxaliplatin both in blood and peritoneal fluid.

SECONDARY OBJECTIVES:

I. Determine tumor-cell intrinsic effects, modulation of the tumor immune microenvironment, and changes in the makeup of circulating immune cells in response to IP 5FU+oxaliplatin.

II. Identify preliminary response from IP 5FU+oxaliplatin: assess the rate of conversion from unresectable to resectable (determined by peritoneal carcinomatosis index [PCI] decreasing to < 20) and response rates by imaging criteria.

OUTLINE: This is a dose-escalation study of 5FU and oxaliplatin followed by a dose-expansion study.

Patients undergo placement of indwelling IP port for chemotherapy infusion. Patients receive oxaliplatin and 5FU over 1-2 hours via IP infusion on days 1 and 15 of each cycle. Cycles repeat every 4 weeks for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo diagnostic laparoscopy, biopsy, computed tomography (CT)/magnetic resonance imaging (MRI), and collection of blood samples at screening and on study and undergo collection of IP fluid samples on study.

After completion of study treatment, patients are followed up for 30 days. Patients with confirmed disease progression or who start a new anti-cancer therapy are followed up every 12 weeks until death, withdrawal of consent, or end of study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Biopsy proven colorectal cancer with peritoneal metastasis. Patients with extraperitoneal metastases will not be eligible. Patients with involvement of intra-abdominal lymph nodes may be eligible at the discretion of the treating physician
* Primary colorectal cancer may either be left in place or have been resected prior to study enrollment
* Patients are allowed to have received prior colorectal cancer-directed systemic therapy.
* Not previously undergone cytoreductive surgery and hyperthermic intraperitoneal chemotherapy (HIPEC) for colorectal cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 at the time of enrollment
* Absolute neutrophil count (ANC) ≥ 1,500 /mcL
* Platelets ≥ 100,000 / mcL
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance ≥ 60 mL/min for patient with creatinine levels > 1.5 x institutional ULN (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl])

  * Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ ULN for patient with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN

  * Both values must be in the specified range
* Albumin >= 2.5 g/dL
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Patients on anticoagulation or antiplatelet agents may be enrolled at the discretion of the treating physician, provided these can be safely held as needed for surgical procedures
* Anticipated life expectancy of ≥ 6 months
* Willing to comply with study procedures
* Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study and at least 9 months after the last dose of study medication
* For female patients of childbearing potential, a negative pregnancy test is required at or within 7 days prior to enrollment
* Be willing and able to understand and sign the written informed consent document
* Be willing to undergo two diagnostic laparoscopies with tumor biopsy tissue. Patients must consent to on-treatment biopsies prior to initiation of clinical trial
* Be willing to provide peripheral blood and peritoneal samples for correlative studies

Exclusion Criteria:

* Patients who are receiving any other investigational drugs
* Evidence of metastatic disease other than peritoneum based on standard of care (SOC) imaging
* Patients with primary mucinous appendiceal tumors will not be eligible. These tumors often produce mucin, which may affect the penetration of IP chemotherapy. Patients with non-mucinous appendiceal adenocarcinomas will be eligible.
* Patients with >= grade 2 peripheral neuropathy
* Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, cardiac arrhythmia, active bleeding diatheses, and psychiatric illness/social situations that would limit compliance with study requirements
* Major surgical procedure or significant traumatic injury less than 3 weeks or those who receive minor surgical procedures within 1 week from first dose of study drug administration
* Known active chronic infections - uncontrolled human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome (AIDS), known active (i.e., with detectable polymerase chain reaction [PCR]) hepatitis B or C
* Cirrhosis (Child-Pugh B or worse) or cirrhosis with history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis
* Pregnancy or breastfeeding
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 1 year
  MTD will be determined based on isotonic regression. Specifically, the MTD will be selected as the dose for which the isotonic estimate of the toxicity rate is closest to the targeted dose limiting toxicities via Bayesian optimal interval software.
Incidence of adverse events | Up to 30 days after completion of study treatment
  Adverse events (AEs) will be classified and attributed using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 and will be summarized within and across dose levels using descriptive statistics. The overall number and percentage of patients experiencing AEs and toxicities will be summarized and reported as across all event types. All patients who have received at least one dose of the therapeutic agents will be evaluable for toxicity and tolerability.
Area under the curve | At the end of Cycle 1 (each cycle is 28 days)
  Will be computed using non-compartmental and compartmental methods. Will use graphical analyses as well as repeated measure models (linear or nonlinear mixed models, generalized estimating equations) to assess the pharmacokinetic markers in relation to clinical treatment outcomes, recognizing some inherent limitations due to sample size.
Clearance | At the end of Cycle 1 (each cycle is 28 days)
  Will be computed using non-compartmental and compartmental methods. Will use graphical analyses as well as repeated measure models (linear or nonlinear mixed models, generalized estimating equations) to assess the pharmacokinetic markers in relation to clinical treatment outcomes, recognizing some inherent limitations due to sample size.
Volume of distribution | At the end of Cycle 1 (each cycle is 28 days)
  Will be computed using non-compartmental and compartmental methods. Will use graphical analyses as well as repeated measure models (linear or nonlinear mixed models, generalized estimating equations) to assess the pharmacokinetic markers in relation to clinical treatment outcomes, recognizing some inherent limitations due to sample size.
Half-life | At the end of Cycle 1 (each cycle is 28 days)
  Will be computed using non-compartmental and compartmental methods. Will use graphical analyses as well as repeated measure models (linear or nonlinear mixed models, generalized estimating equations) to assess the pharmacokinetic markers in relation to clinical treatment outcomes, recognizing some inherent limitations due to sample size.

SECONDARY OUTCOMES:
Tumor-cell intrinsic effects in response to IP 5FU+oxaliplatin | Up to 16 weeks
  Samples obtained from baseline and after 4 cycles will be studied. Data collected will be descriptive and exploratory, and provide limited estimates of variability given the small sample sizes at each dose level. Results will be summarized using descriptive statistics (i.e., means, standard deviations, 95% confidence intervals for continuous variables, and frequencies for discrete data.
Modulation of the tumor microenvironment in response to IP 5FU+oxaliplatin | Up to 16 weeks
  Samples obtained from baseline and after 4 cycles will be studied. Data collected will be descriptive and exploratory, and provide limited estimates of variability given the small sample sizes at each dose level. Results will be summarized using descriptive statistics (i.e., means, standard deviations, 95% confidence intervals for continuous variables, and frequencies for discrete data.
Changes in the makeup of circulating immune cells in response to IP 5FU+oxaliplatin | Up to 16 weeks
  Samples obtained from baseline and after 4 cycles will be studied. Data collected will be descriptive and exploratory, and provide limited estimates of variability given the small sample sizes at each dose level. Results will be summarized using descriptive statistics (i.e., means, standard deviations, 95% confidence intervals for continuous variables, and frequencies for discrete data.
Rate of conversion from unresectable to resectable | At time of second laparoscopy, after 4 cycles of treatment (16 weeks)
  Resectable disease will be determined by peritoneal carcinomatosis index decreasing to < 20. Will be summarized and 95% exact binomial confidence interval will be provided.
Overall response rate | Up to 16 weeks
  Will be evaluated using imaging criteria. Overall response rate (partial response + complete response) will be summarized and 95% exact binomial confidence interval will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Arjun Mittra, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - UT Southwestern/Simmons Cancer Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu